CLINICAL TRIAL: NCT02713841
Title: Samba-01: A Phase 1/2 Trial Investigating the Pharmacokinetics, Pharmacodynamics and Safety of Inhaled Insulin in Subjects With Type 1 Diabetes
Brief Title: Pharmacologic Response and Safety of Inhaled Insulin in Type 1 Diabetes
Acronym: Samba-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dance Biopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Samba-01
Record Dates: First submitted 2016-03-02; First posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Inhaled insulin (LOM) (Experimental): single 50 unit dose of Dance inhaled insulin administered using the Adagio-01 inhaler device with a low output mesh (aerosol particles sized 3.5-4.0 μm)
  Interventions: Drug: inhaled human insulin (INH)
- Inhaled insulin (MOM1) (Experimental): single 50 unit dose of Dance inhaled insulin administered using the Adagio-01 inhaler device with a medium output mesh (aerosol particles sized 4.3-4.8 μm)
  Interventions: Drug: inhaled human insulin (INH)
- Inhaled insulin (MOM2) (Experimental): repeat of single 50 unit dose of Dance inhaled insulin administered using the Adagio-01 inhaler device with a medium output mesh (aerosol particles sized 4.3-4.8 μm)
  Interventions: Drug: inhaled human insulin (INH)
- Inhaled insulin (HOM) (Experimental): single 50 unit dose of Dance inhaled insulin administered using the Adagio-01 inhaler device with a high output mesh (aerosol particles sized 5.0-5.5 μm)
  Interventions: Drug: inhaled human insulin (INH)
- subcutaneous insulin lispro (LIS) (Active Comparator): single 6 unit dose of insulin lispro administered subcutaneously
  Interventions: Drug: sc insulin lispro (LIS)

INTERVENTIONS:
Drug: inhaled human insulin (INH) — recombinant human insulin administered with Adagio-01 inhaler device
  Other Names: Dance-501
  Arms: Inhaled insulin (HOM); Inhaled insulin (LOM); Inhaled insulin (MOM1); Inhaled insulin (MOM2)
Drug: sc insulin lispro (LIS) — insulin lispro administered subcutaneously
  Arms: subcutaneous insulin lispro (LIS)

SUMMARY:
The purpose of this study was to compare the pharmacokinetic (PK) response after inhaled insulin administration with 3 different inhalation regimens and with subcutaneous insulin administration.

DETAILED DESCRIPTION:
This first-in-human trial investigated the optimal particle size for absorption of Dance-501, an aerosolized liquid human insulin for inhalation (INH).

Twelve subjects with type 1 diabetes received an INH dose (50 IU) using an inhaler on 4 visits and 6 U insulin lispro (LIS) sc on a separate visit to assess relative bioavailability (FREL) of INH. The inhaler was configured to generate insulin aerosol particles sized 3.5-4.0 μm (low output mesh; LOM), 4.3-4.8 μm (medium output mesh; MOM) or 5.0-5.5 μm (high output mesh; HOM) during low inspiratory flow. To assess within subject variability, MOM was used twice. Pharmacokinetics (PK) were measured up to 8 hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus treated with multiple daily insulin injections or continuous subcutaneous insulin infusion and total daily insulin dose less than 1.2 units/kg/day.
* Body mass index 18.0 - 28.0 kg/m2.
* Hemoglobin A1c less than or equal to 9%.
* Forced vital capacity and forced expiratory volume in one second at least 75% of predicted normal values for race, age, gender and height.
* Fasting C-peptide less than 0.3 nmol/L.

Exclusion Criteria:

* Subjects with any condition possibly affecting drug absorption from the lung, in particular subjects with decreased lung function or subjects taking bronchodilators or subjects who smoke.
* Active or chronic pulmonary disease.
* Any clinically significant major disorders other than diabetes mellitus.
* Decompensated heart failure at any time or angina pectoris within the last 12 months or acute myocardial infarction at any time.
* Proliferative retinopathy or severe neuropathy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Area under the insulin human / insulin lispro concentration-time curve from 0 to 8 hours (AUCINS,0-8h) | 0 to 8 hours
Bioavailability | 0 to 8 hours
  Relative delivery efficiency (FREL) of inhaled human insulin (INH) compared to s.c. injected insulin lispro (LIS)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH

IPD SHARING:
Plan to Share IPD: No